CLINICAL TRIAL: NCT06602765
Title: Comparative Analysis of Interventions for Prevention of Dental Caries in School Children: A Randomized Controlled Trial
Brief Title: Comparative Analysis of Interventions for Prevention of Dental Caries in School Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Kulsoom Rizvi, Professor, Bahria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BUHS-IRB#061/24
Record Dates: First submitted 2024-07-21; First posted 2024-09-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Prevention of Dental Caries
Keywords: Fissure sealant; Fluoride; Caries; Saliva; Dietary counselling
MeSH Terms: interventions — Toothbrushing

STUDY DESIGN:
Intervention Model Description: Control, Interventional group 1, Interventional group 2
Who Masked: Outcomes Assessor
Masking Description: A single-blind trial will be conducted where the outcome assessor/statistician will be blind to the intervention received by the participants in different groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tooth-brushing (Active Comparator): In Control arm, tooth brushing with fluoride toothpaste using pea-sized toothpaste, using bass technique.
  Interventions: Other: Tooth brushing, tooth paste containing 1450ppm fluoride
- tooth-brushing and dietary counselling (Active Comparator): In intervention arm 1, tooth brushing with fluoride toothpaste using pea-sized toothpaste, using the bass technique, and dietary counselling.
  Interventions: Other: Tooth brushing, tooth paste containing 1450ppm fluoride
- tooth-brushing , dietary counselling and fissure sealing of 1st permanent molar (Active Comparator): In the intervention arm 2, tooth brushing with fluoride toothpaste using pea-sized toothpaste, using the bass technique, dietary counseling, and application of fissure sealant on a permanent first molar.
  Interventions: Other: Tooth brushing, tooth paste containing 1450ppm fluoride

INTERVENTIONS:
Other: Tooth brushing, tooth paste containing 1450ppm fluoride — brushing with fluoride toothpaste, dietary counselling for caries prevention and application of fissure sealant compound on first permanent t molars.
  Other Names: dietary counselling; fissure sealent, Glassionomer cement

SUMMARY:
A study aims to assess the most effective preventive interventions to address the widespread issue of dental caries, affecting an estimated 2 billion people in permanent teeth and over 500 million children in primary teeth globally. Notably, in Pakistan, over 90% of caries-affected teeth are untreated. Despite schools being a platform for public health initiatives, there is limited evidence on oral health promotion in low and middle-income countries. This study compares different preventive strategies' effectiveness and cost-efficiency for caries prevention in schoolchildren.

The randomized controlled trial will occur in Naval Schools of Karachi under the Pakistan Navy Educational Trust (PNET) over one year, including intervention and follow-up periods. The interventions include a combination of fluoride toothpaste, dietary counselling, and fissure sealant application. A multi-stage sampling method will select schools and classes, while convenience random sampling will select 180 children for the study. A single-blind trial will be conducted, with the data analyst unaware of the intervention groups.

Participants will be divided into three groups. Group 1 (Control) will use fluoride toothpaste and be instructed to brush twice daily. Group 2 (Intervention-1) will receive 14500 ppm fluoride toothpaste and oral health education. Group 3 (Intervention-2) will include the treatments from Group 2 plus fissure sealants on the first permanent molars. Parents in Groups 2 and 3 will receive a standardized advice sheet to reinforce oral hygiene practices at home.

The study will collect baseline demographic data, including age, gender, socioeconomic status, family education, existing oral hygiene practices, dental knowledge, and dentition status. Oral examinations will be conducted according to international standards. Statistical analysis will employ Chi-Square, ANOVA, and logistic regression tests, with a significance level set at 0.05.

The study aims to determine the most effective preventive strategy by comparing the reduction in dental caries incidence across the groups. The findings will guide recommendations for implementing the most effective intervention on a larger scale in schools, with the goal of reducing the burden of dental caries in children.

DETAILED DESCRIPTION:
Ethical Approval approved by the BUHSC ethical committee. School administrations will be approached for permission. Consent forms will be sent to the parents of the children before the data collection visit. The data collection team comprised of 06 members will visit the selected schools. A signed consent form will be taken, and verbal consent will be obtained from the children as well. The children fulfilling the inclusion criteria will be sequenced as a list. Randomization will be done through SNOSE - a sequential number of opaque sealed envelopes will be done, and the students will then be allocated in 3 groups.

PI, Co-PI, and 05 team members will conduct oral examinations in the selected schoolyard or inside a classroom, following the standard international guidelines (WHO 2013). In addition, the baseline demographic data will also be collected comprising of age, gender, socioeconomic status (SES), family education and existing oral hygiene practices, dental knowledge, and dentition status by the parents and participants. Group 1 (Control) will be given fluoride toothpaste containing 1450 ppm Fluoride and will be asked to brush at least twice daily with a pea-sized amount of toothpaste, using the modified bass technique. This will be considered as control. Some intervention in the control group will also address the ethical issues. Parents will be guided for the tooth brushing.

Group 2 (Intervention -1) will be given fluoride toothpaste containing 1450 ppm Fluoride and will be asked to brush at least twice daily with a pea-sized amount of toothpaste and oral health education. A modified bass technique for tooth brushing will be used. Oral health education through audio-visual aids, pamphlets, and live demonstrations on study models will cover proper tooth brushing techniques, the use of a good toothbrush, and healthy eating habits, including special emphasis on proteins and dairy products and alternate use of sugars in daily routine. E.g. soft drinks that are high in sugar can be replaced with drinking milk and water.

Group 3 (Intervention -1) will be given fissure sealants on 1st permanent molar along with the strategy given to Group 2. Fissure sealing compounds, Glass ionomer will be used on school children who will qualify for inclusion criteria. Mobile Dental Unit and fissure sealant kit will be taken to the site and children will be provided fissure sealant in their setting.

In the intervention group (2 and 3) parents will also be given an Evidence-Based standardized parental advice sheet to reinforce instructions at home.

The saliva of school children will be collected by spitting in a test tube. For children over the age of 6, saliva can be collected using the expectoration, or spit method. In this process, the child is instructed to keep their mouth closed for three minutes without swallowing, allowing saliva to accumulate before spitting it into a collection tube. However, some children may struggle with this technique due to the challenge of not swallowing for an extended period. An alternative method is the drainage technique. Here, the child is first asked to swallow their saliva to stimulate the production of more saliva. Then, with their lips slightly parted, the saliva is allowed to drain directly into the collection tube The samples will be taken to the laboratory within 02 hours of collection Streptococcus mutans count will be conducted on collected saliva at the first visit to provide an initial bacterial count as baseline data before intervention and after six-month and 12-month bacterial count after the intervention. The primary medium used to identify streptococci is Mitis-Salivarius agar or its variant with bacitracin (MSB). Additionally, saliva's pH, flow rate, and buffering capacity will be measured in the lab. The first visit will be followed by six months and 12 months respectively. A preliminary pilot study will be undertaken with a limited sample size to assess the practicality of the interventions and enhance the process of collecting data.

The data collected through the questionnaire and log book filled by parents at home will be computerized, followed by converting it into the appropriate SPSS files. The outcome variables for assessing dental caries will be measured by ICDAS. The ICDAS is a two-digit coding method. One for caries and the other for sealant and restorations. In this research, only the caries coding method will be used. For caries, the method ranges from sound teeth (code 0), through enamel caries lesions (codes 1-3), to carious lesions in dentine (codes 4-6). For sealant and restoration, the method ranges from 0 to 8 as follows: 0 = Sound, 1 = Sealant, partial, 2 = Sealant, full, 3 = Tooth-coloured restoration, 4 = Amalgam restoration, 5 = Stainless steel crown, 6 = Porcelain or gold or Porcelain-Fused-to-Metal (PFM) crown or veneer, 7 = Lost or broken restoration, 8 = Temporary restoration (will not be used). Caries Codes (0 = sound tooth surface; A = first visual change in enamel; B = distinct visual change in enamel; 3 = enamel breakdown, no dentine visible; 4 = dentinal shadow (not cavitated into dentine); 5 = distinct cavity with visible dentine; 6 = extensive distinct cavity with visible dentine); Missing Teeth (97 = extracted due to caries; 98 = missing for other reasons; 99 = un-erupted).

Salivary indicators i.e. salivary flux - 0.3-0.4 ml/min. Salivary pH - 5-5.8, high acidity; 6.0-6.6, moderate acidity; 6.8-7.8, normal salivary pH Salivary buffer capacity - 3-30 mg/100 ml. Salivary Mutans count - < 10^5 CFU/ml saliva or ≥ 10^5 CFU/ml saliva. The study will use the CONSORT checklist for reporting the randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

Schoolchildren aged 6-7 years Sound 1st permanent molars Consent obtained from parents/guardians Cooperative Children

Exclusion Criteria:

1st Permanent molar has not erupted. Children with disability. Special Children (e.g. Down syndrome)

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-10-05 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevention of dental Caries | 1 year
  Compare the effectiveness of the combination of different preventive strategies which include tooth brushing with fluoride toothpaste, dietary counselling, and fissure sealant application for reducing the incidence of dental caries among school children

SECONDARY OUTCOMES:
Dietary Analysis | 1 year
  Dietary analysis to understand the risk factors and mechanisms underlying dental caries development among school children
Streptococcus mutans in Saliva | 1 year
  Determine the contribution of saliva tests for Streptococcus mutans presence

CONTACTS AND LOCATIONS:
Overall Officials: Kulsoom F Rizvi, MSc, Principal Investigator — Bahria University
Locations (1):
- Pakistan Navy Educational Trust, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No